CLINICAL TRIAL: NCT04310527
Title: A Phase 1, Open-label, Single-Center, Randomized, Three-period, Two-Sequence Crossover Study to Assess Relative Bioavailability of Enasidenib (CC-90007) Sprinkle Formulation Relative to the Reference Tablet Formulation and to Assess the Effect of Food on the Pharmacokinetics of Sprinkle Formulation in Healthy Adult SubjectsHEALTHY ADULT SUBJECTS
Brief Title: Bioavailability of Enasidenib (CC-90007) Sprinkle Formulation Relative to the Reference Tablet Formulation and Effect of Food on the Pharmacokinetics of Sprinkle Formulation in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC-90007-CP-006; U1111-1243-9124 (Registry Identifier: WHO)
Expanded Access: NCT03723057 (No longer available)
Record Dates: First submitted 2020-03-04; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers
Keywords: Enasidenib; CC-90007; pharmacokinetics; Healthy Adults
MeSH Terms: interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A: Administration of enasidenib fasted (Experimental): A single oral 100 mg dose of enasidenib reference formulation will be given under fasted condition.
  Interventions: Drug: Enasidenib
- Treatment B: Administration of enasidenib fasted (Experimental): A single oral 100 mg dose of enasidenib test formulation will be given under fasted condition.
  Interventions: Drug: Enasidenib
- Treatment C: Administration of ensidenib fed (Experimental): A single oral 100 mg dose of enasidenib test formulation will be given under fed condition.
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — Enasidenib

SUMMARY:
This is an open-label, single-center, randomized, three-period, two-sequence crossover study in healthy adult subjects to occur at one site in the United States. This study will evaluate the relative Bioavailability (BA) of an enasidenib sprinkle formulation, compared to the reference tablet formulation, when taken in the fasted state. This study will also evaluate the Pharmacokinetics (PK) of the enasidenib sprinkle formulation after a single oral dose in the fed state to assess the food effect. The study will consist of a Screening phase, a Treatment phase, and a Follow-up phone call. Approximately 28 healthy adult subjects (males or non-pregnant females) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must understand and voluntarily sign an Informed Consent Form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
3. Subject is male, or non-pregnant and non-nursing female ≥ 18 and ≤ 55 years of age at the time of signing the ICF.
4. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before Screening, or be postmenopausal (defined as 24 consecutive months without menses before Screening, with a follicle-stimulating hormone [FSH] level of > 40 IU/L at Screening).
5. Females of childbearing potential (FCBP)1 may participate, providing they meet the following conditions:

   • Agree to practice true abstinence2 from sexual intercourse or to use highly effective contraceptive methods (eg, combined [containing estrogen and progestogen] or progestogen-only associated with inhibition of ovulation, oral, injectable, intravaginal ring (e.g. vaginal hormonal ring), patch, or implantable hormonal contraceptive; bilateral tubal occlusion; intra-uterine device; intrauterine hormone-releasing system; or male partner sterilization [note that vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the Females of childbearing potential (FCBP) trial participant and that the vasectomized partner has received medical assessment of the surgical success]) at screening and throughout the study, and for 2 months following the last study treatment;

   • Have a negative serum β-subunit of human chorionic gonadotropin (β-hCG) pregnancy test (sensitivity of at least 25 mIU/mL) at Screening; and

   • Have a negative serum β-hCG pregnancy test (sensitivity of at least 25 mIU/mL) within 72 hours prior to the start of study treatment in the Treatment Phase (note that the screening serum pregnancy test can be used as the test prior to the start of study treatment in the Treatment Phase if it is performed within the 72-hour timeframe).
6. Male subjects must:

   a. Practice true abstinence3 (which must be reviewed on a monthly basis and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or FCBP while participating in the study and for at least 2 months after the last dose of Investigational product (IP), even if he has undergone a successful vasectomy.
7. Subject has body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at Screening.
8. Subject has a satisfactory medical assessment with no clinically significant or relevant abnormalities determined by medical history, PE, vital signs, 12-lead ECG, and clinical laboratory evaluation (hematology, clinical chemistry, and urinalysis) that are reasonably likely to interfere with the subject's participation in, or ability to complete the study as assessed by the Investigator.

   a. Subject vital signs are as follows:

   - Tympanic body temperature:35.0 - 37.5°C.

   - Supine blood pressure (BP) after at least 5 minutes supine rest: i. Systolic BP: 90 - 140 mmHg ii. Diastolic BP: 40 - 90 mmHg b. Supine heart rate (after at least 5 minutes of rest):

   - 45 - 90 beats per minute (measured during vital sign assessment)

   - Subject has a normal or clinically acceptable 12-lead ECG at Screening.

In addition:

i. If male, subject has a QT interval corrected for heart rate using Fridericia's formula (QTcF) value ≤ 430 msec at Screening. ii. If female, subject has a QTcF value ≤ 450 msec at Screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness as determined by medical history, Physical examination (PE), vital signs, 12-lead Electrocardiogram (ECG), and clinical laboratory evaluation (hematology, clinical chemistry, and urinalysis) that would place the subject at unacceptable risk or prevent the subject from participating in the study.
2. Subject has any condition that confounds the ability to interpret data from the study.
3. Subject has a history of multiple (ie, 2 or more) or severe drug allergies.
4. Subject has been:

   1. previously exposed to enasidenib or;
   2. has been exposed to an investigational drug (new chemical entity) within 90 days preceding the first dose administration, or five half-lives of that investigational drug, if known (whichever is longer).
5. Subject has used any prescription drugs or over-the-counter medication (including multi-vitamins) except those permitted in within 14 days prior to Day 1.
6. Subject has consumed herbal remedies or dietary supplements containing St. John's Wort, in the 3 weeks before Day 1.
7. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion.

   1. Chronic or permanent conditions such as bariatric procedures, extensive bowel resections, irritable bowel syndrome, etc. are exclusionary at any time prior to Screening.
   2. Acute conditions such as dysentery or acute gastroenteritis are exclusionary if they resolved less than 14 days before Screening.
   3. Appendectomy and cholecystectomy are acceptable.
8. Subject has a history of drug or alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before the first dose administration, or positive Screening or Day -1 test reflecting consumption of illicit drugs or alcohol.
9. Subject is known to have any viral hepatitis infection (including carrier state) or has a positive result to the tests for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV) antibodies at Screening.
10. Subject smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
11. Subject is part of the clinical staff personnel or a family member of the clinical site staff.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | UP to approximately 14 days
  Observed maximum concentration
Pharmacokinetics - AUC0-∞ | UP to approximately 14 days
  Area under the concentration-time curve calculated from time zero to infinity
Pharmacokinetics - AUC0-t | UP to approximately 14 days
  Area under the concentration-time curve calculated from time zero to the last measured time point
Pharmacokinetics - Tmax | UP to approximately 14 days
  Time to Cmax
Pharmacokinetics - t½ | UP to approximately 14 days
  Terminal elimination half-life
Pharmacokinetics - CL/F | UP to approximately 14 days
  Apparent clearance of drug from plasma after extravascular administration
Pharmacokinetics - Vz/F | UP to approximately 14 days
  Apparent volume of distribution during the terminal phase

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene
Locations (1):
- PPD Development, LP, Austin, Texas, United States